CLINICAL TRIAL: NCT03960580
Title: A 24-Week Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study Evaluating the Efficacy and Safety of Intranasal Administration of 186 and 372 μg of OPN-375 Twice a Day (BID) in Subjects With Chronic Rhinosinusitis Without the Presence of Nasal Polyps
Brief Title: Study Evaluating the Efficacy and Safety of Intranasal Administration of OPN-375 in Subjects With Chronic Rhinosinusitis Without the Presence of Nasal Polyps
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Optinose US Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPN-FLU-CS-3206
Record Dates: First submitted 2019-05-20; First posted 2019-05-23 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Chronic Rhinosinusitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OPN-375 186 μg BID (Active Comparator): OPN-375 186 μg BID x 24 Weeks
  Interventions: Drug: OPN-375
- OPN-375 372 μg BID (Active Comparator): OPN-375 372 μg BID x 24 Weeks
  Interventions: Drug: OPN-375
- Placebo (Placebo Comparator): Matching Placebo BID x 24 Weeks
  Interventions: Drug: OPN-375

INTERVENTIONS:
Drug: OPN-375 — OPN-375, BID

SUMMARY:
This is a 24-week randomized, double-blind, placebo-controlled, parallel-group, multicenter study to evaluate the efficacy and safety of intranasal administration of 186 and 372 μg twice daily (BID) of OPN-375 in subjects with chronic Rhinosinusitis (CRS) without nasal polyps

DETAILED DESCRIPTION:
The primary objective of this study is to compare the efficacy of intranasal administration of twice-daily doses of 186 and 372 µg of OPN-375 (fluticasone propionate) with placebo in subjects with chronic rhinosinusitis using the following co-primary endpoints:

1. A change from baseline in symptoms as measured by the average morning composite score of nasal congestion, facial pain or pressure sensation, and nasal discharge (anterior and/or posterior) at the end of Week 4.
2. A change from baseline to Week 24/Early Termination (ET) in the average percent of the volume opacified in the ethmoid and maxillary sinuses.

ELIGIBILITY:
Inclusion Criteria:

1. men or women aged 18 years and older at baseline visit
2. women of child bearing potential must be abstinent, or if sexually active,

   1. be practicing an effective method of birth control (eg, prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method [eg, condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel], or male partner sterilization) before entry and throughout the study, or
   2. be surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), or
   3. be postmenopausal (amenorrhea for at least 1 year)
3. women of child-bearing potential must have a negative urine pregnancy test at Visit 1 (Screening)
4. must have a history of chronic sinusitis and be currently experiencing 2 or more of the following symptoms, 1 of which has to be either nasal congestion or nasal discharge (anterior and/or posterior nasal discharge) for equal to or greater than 12 weeks:

   * nasal congestion
   * nasal discharge (anterior and/or posterior nasal discharge)
   * facial pain or pressure
   * reduction or loss of smell
5. endoscopic evidence of nasal mucosal disease, with edema or purulent discharge; or polyps/polypoid tissue <Grade 1 in middle meatus, bilaterally
6. must have confirmatory evidence via a computed tomography(CT) scan of bilateral sinus disease (have at least 1 sinus on each side of nose with a Lund-Mackay score of ≥1)
7. baseline CT scan must show a combined ≥25% opacification of the ethmoid sinuses and ≥25% opacification of at least 1 maxillary sinus
8. must have at least moderate symptoms (as defined in protocol) of nasal congestion as reported by the subject, on average, for the 7-day period preceding Visit 1 (Screening) run-in
9. must have an average morning score of at least 1.5 for congestion on the Nasal Symptom Scale (as defined in protocol) recorded on the subject diary over a 7-day period during the first 14 days of the single-blind run-in period
10. must demonstrate an ability to correctly complete the daily diary during the run-in period to be eligible for randomization
11. Subjects with comorbid asthma or chronic obstructive pulmonary disorder (COPD) must be stable with no exacerbations (eg, no emergency room visits, hospitalizations, or oral or parenteral steroid use) within the 3 months before Visit 1 (Screening). Inhaled corticosteroid use must be limited to stable doses of no more than 1,000 μg/day of beclomethasone (or equivalent) for at least 3 months before Visit 1 (Screening) with plans to continue use throughout the study.
12. Subjects with aspirin-exacerbated respiratory disease, who have undergone aspirin desensitization and are receiving daily aspirin therapy, must be receiving therapy for at least 6 months prior to Visit 1.
13. must be able to cease treatment with intranasal steroids, inhaled corticosteroids (except permitted doses listed above for asthma and COPD) at the screening visit.
14. must be able to cease treatment with oral and nasal decongestants and antihistamines at Visit 1 (Screening)
15. must be able to use the exhalation delivery system correctly; all subjects will be required to demonstrate correct use with the practice exhalation delivery system (EDS) at Visit 1 (Screening).
16. must be capable, in the opinion of the investigator, of providing informed consent to participate in the study. Subjects must sign an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

1. women who are pregnant or lactating
2. inability to have each nasal cavity examined for any reason, including nasal septum deviation
3. inability to achieve bilateral nasal airflow
4. is currently taking XHANCE®
5. have previously used XHANCE® for more than 1 month and did not achieve an adequate symptomatic response
6. the nasal/sinus anatomy prevents the accurate assessment of sinus volume via CT scan
7. history of sinus or nasal surgery within 6 months before Visit 1 or has not healed from a prior sinus or nasal surgery
8. have current evidence of odontogenic sinusitis, sinus mucocele (the affected sinus is completely opacified and either the margins are expanded and/or thinned OR there are areas of complete bone resorption resulting in bony defect and extension of the "mass" into adjacent tissues), evidence of allergic fungal sinusitis, or evidence of complicated sinus disease (including, but not limited to, extension of inflammation outside of the sinuses and nasal cavity)
9. have a paranasal sinus or nasal tumor
10. have polyp grade ≥1 (polyp that is free on 5 sides and has a stalk) on either side of the nose as determined by the nasoendoscopy at screening
11. have a nasal septum perforation
12. have had more than 1 episode of epistaxis with frank bleeding in the month before Visit 1 (Screening)
13. have evidence of significant mucosal injury, ulceration (eg, exposed cartilage) on Visit 1 (Screening) nasal examination/nasoendoscopy
14. have current, ongoing rhinitis medicamentosa (rebound rhinitis)
15. have significant oral structural abnormalities (eg, a cleft palate)
16. have a diagnosis of cystic fibrosis
17. history of Churg-Strauss syndrome or dyskinetic ciliary syndromes
18. symptom resolution or last dose of antibiotics for purulent nasal infection, acute sinusitis, or upper respiratory tract infection has not occurred before Visit 1 or was less than 4 weeks before the CT scan. Potential subjects presenting with any of these infections may be rescreened 4 weeks after symptom resolution.
19. planned sinonasal surgery during the period of the study
20. allergy, hypersensitivity, or contraindication to corticosteroids or steroids
21. has used oral steroids in the past for treatment of chronic sinusitis and did not experience any relief of symptoms
22. has a steroid eluting sinus stent still in place within 30 days of Visit 1
23. allergy or hypersensitivity to any excipients in study drug
24. exposure to any glucocorticoid treatment with potential for systemic effects (eg, oral, parenteral, intraarticular, or epidural steroids, high dose topical steroids) within 1 month before Visit 1 (Screening); except as noted in inclusion criteria for subjects with comorbid asthma or COPD
25. have nasal candidiasis
26. history or current diagnosis of any form of glaucoma or ocular hypertension
27. history of intraocular pressure elevation on any form of steroid therapy
28. history or current diagnosis of the presence (in either eye) of a subcapsular cataract
29. history of immunodeficiency
30. any serious or unstable concurrent disease, psychiatric disorder, or any significant condition that, in the opinion of the investigator could confound the results of the study or could interfere with the subject's participation or compliance in the study
31. have a positive drug screen or a recent (within 1 year of Visit 1 [Screening]) history of drug or alcohol abuse, or dependence that, in the opinion of the investigator could interfere with the subject's participation or compliance in the study
32. have participated in an investigational drug clinical trial within 30 days of Visit 1 (Screening)
33. have received mepolizumab (Nucala®), reslizumab (Cinquair®), dupilumab (Dupixent®), omalizumab (Xolair®), or benralizumab (Fasenra™) within 6 months of Visit 1 (Screening)
34. is using strong cytochrome P450 3A4 (CYP3A4) inhibitors (eg, ritonavir, atazanavir, clarithromycin, indinavir, itraconazole, nefazodone, nelfinavir, saquinavir, ketoconazole, telithromycin, conivaptan, lopinavir, voriconazole)
35. is an employee of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, or is a family member of the employee or the investigator.
36. patients who report unexplained worsening of vision within the past 3 months (e.g. difficulty reading or seeing traffic signs from a distance). A diagnosis of presbyopia established by an eye care professional is not exclusionary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Carothers, Study Director — Optinose US Inc.; John Messina, Study Chair — Optinose US Inc.
Locations (87):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Sacramento Ear, Nose & Throat Surgical and Medical Group Inc, Folsom, California
  - BioSolutions Clinical Research Center, La Mesa, California
  - Veterans Administration Greater Los Angeles Healthcare System, Los Angeles, California
  - Sacramento Ear, Nose & Throat Surgical and Medical Group, Roseville, California
  - Asthma and Allergy Associates, Colorado Springs, Colorado
  - Sher Allergy Specialists, Largo, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - Best Clinical Trials, New Orleans, Louisiana
  - University of Missouri, Dept of Otorlaryngology, Columbia, Missouri
  - Mount Sinai Downtown Union Square, New York, New York
  - Northwell Health at ENT and Allergy Associates, New York, New York
  - Charlotte Eye Ear Nose and Throat Assoc., PA, Matthews, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - ENT & Allergy Partners, LLC, Summerville, South Carolina
  - Pasha Snoring & Sinus Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Allergy, Asthma & Sinus Center, SC, Greenfield, Wisconsin
- Australia (8):
  - Otopure Pty Ltd, Bella Vista, New South Wales
  - Vale Medical Practice, Brookvale, New South Wales
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Browns Plains Family Practice, Browns Plains, Queensland
  - Casey Superclinic, Berwick, Victoria
  - Camberwell Road Medical Practice, Hawthorn East, Victoria
  - Mirrabooka Medical Centre, Mirrabooka, Western Australia
  - Latitude Clinical Research, Spearwood, Western Australia
- Bulgaria (9):
  - UMHAT Kaspela EOOD, Plovdiv
  - Medical Center Iskar EOOD, Sofia
  - MHAT Serdika EOOD, Sofia
  - MC N.I. Pirogov EOOD, Sofia
  - MHAT - Central Clinical Base Sofia Medical Institute Ministry of Interior, Sofia
  - MMA MHAT - Sofia, Sofia
  - DCC Convex EOOD, Sofia
  - MHAT Trakiya EOOD, Stara Zagora
  - DCC "Mladost - M Varna" OOD, Varna
- Czechia (7):
  - Nemocnice Rudolfa a Stefanie Benesov, a.s., ORL oddeleni, Benešov
  - FN Hradec Kralove, Klinika ORL, Hradec Králové
  - Pro-audio s.r.o., Mladá Boleslav
  - MUDr. Pavel Navratil, ORL ambulance, Olomouc
  - Nemocnice Pardubického kraje - Pardubická nemocnice, Pardubice
  - VFN v Praze, oddeleni ORL, Prague
  - AXON Clinical s.r.o., Prague
- Georgia (7):
  - Ltd Acad. Fridon Todua Medical Center- Research, Tbilisi
  - Ltd Israel-Georgian Medical Research Clinic - Helsicore, Tbilisi
  - JSC Curatio, Tbilisi
  - Ltd New Hospitals, Tbilisi
  - Ltd Simon Khechinashvili University Hospital, Tbilisi
  - Ltd Tbilisi Heart Center, Tbilisi
  - Ltd Aversi Clinic, Tbilisi
- New Zealand (4):
  - P3 Research Tauranga Ltd., Tauranga, Bay of Plenty
  - Optimal Clinical Trials, Auckland
  - Clinical Trials New Zealand, Hamilton
  - P3 Research Wellington Ltd., Wellington
- Poland (16):
  - Przychodnia "Narutowicza", Inowrocław, Kuyavian-Pomeranian Voivodeship
  - Indywidualna Specjalistyczna Praktyka Lekarska J. Slifirski, Kęty, Lesser Poland Voivodeship
  - Centrum Medyczne All-Med, Krakow, Lesser Poland Voivodeship
  - ReumaClinic Gabinet Reumatologiczny, Bialystok
  - Centrum Medyczne MedSen Sp. z o.o., Bialystok
  - Centrum Medyczne Kwiatowa, Bydgoszcz
  - Synexus Polska Sp. Z o. o., Oddzial w Gdyni ul. Luzycka 3c, Gdynia
  - Centrum Medyczne Angelius Provita, Katowice
  - Centrum Alergologii Specjalistyczna Przychodnia Alergologiczna, Lublin
  - Centrum Medyczne Lucyna Andrzej Dymek S.C., Strzelce Opolskie
  - NZOZ "Ignis" dr med. Alicja Lobinska, Świdnik
  - NZOZ Przychodnia Medycyny Rodzinnej, Świętochłowice
  - NZOZ Centrum Medyczne LiMED, Tarnowskie Góry
  - Synexus Polska Sp. z.o.o. Oddzial w Warszawie, Warsaw
  - Synexus Polska Sp.zo.o. Oddział we Wrocławiu, Wroclaw
  - Mini-Clinic Paweł Białogłowski, Łańcut
- Romania (6):
  - S.C. Centrul Medical Unirea S.R.L. Brasov, Brasov
  - SC Centrul Medical Unirea srl, Policlinica Primaverii, Bucharest
  - S.C. Euroclinic Hospital S.A., Bucharest
  - Centrul Medical Cardiomed Cluj, Cabinet ORL, Cluj-Napoca
  - Spitalul Clinic Universitar CF Cluj-Napoca, Cluj-Napoca
  - S.C. Centrul Medical Unirea S.R.L - IASI, Campus Medical Iasi - Cabinet ORL, Iași
- Spain (9):
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera, Cadiz
  - Hospital Universitario de Fuenlabrada Servicio de Otorrinolaringología, Fuenlabrada, Madrid
  - Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid
  - Centro Médico Teknon, Barcelona
  - Hospital Universitari Clinic de Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Servicio de Otorrinolaringología, L'Hospitalet de Llobregat
  - Consulta 164 Servicio ORL Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario i Politecnic la Fe, Valencia
- King's Mill Hospital, Sutton in Ashfield, Nottinghamshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching Placebo BID x 24 Weeks
  OPN-375: OPN-375, Twice a Day (BID)
- OPN-375 186 μg BID: OPN-375 186 μg BID x 24 Weeks
  OPN-375: OPN-375, Twice a Day (BID)
- OPN-375 372 μg BID: OPN-375 372 μg BID x 24 Weeks
  OPN-375: OPN-375, Twice a Day (BID)
Period: Overall Study
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Started | 75 | 74 | 74
Completed | 69 | 70 | 71
Not Completed | 6 | 4 | 3
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Marked Randomized in error (patient did not receive study drug) | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID | Total
Number analyzed (Participants) | 75 | 73 | 74 | 222
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 67 | 65 | 63 | 195
  >=65 years | 8 | 8 | 11 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (12.34) | 47.1 (13.75) | 49.4 (13.53) | 48.4 (13.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 40 | 39 | 111
  Male | 43 | 33 | 35 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 74 | 71 | 74 | 219
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 74 | 72 | 73 | 219
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 1 | 0 | 0 | 1
  Romania | 6 | 9 | 9 | 24
  United States | 5 | 5 | 12 | 22
  Czechia | 9 | 4 | 5 | 18
  Poland | 36 | 37 | 30 | 103
  United Kingdom | 0 | 0 | 1 | 1
  Georgia | 7 | 8 | 7 | 22
  Australia | 2 | 1 | 2 | 5
  Bulgaria | 6 | 6 | 4 | 16
  Spain | 3 | 3 | 4 | 10
Intranasal corticosteroid treatment for chronic sinusitis within last 10 years [Number; unit: participants]
  Mometasone furoate | 38 | 28 | 35 | 101
  Fluticasone proprionate | 20 | 15 | 16 | 51
  Fluticasone furoate | 28 | 23 | 24 | 75
  Budesonide | 7 | 3 | 2 | 12
  Beclomethasone | 2 | 2 | 2 | 6
  Triamcinolone | 2 | 2 | 1 | 5
  Fluticasone and azelastine | 14 | 13 | 13 | 40
  Other | 2 | 2 | 2 | 6
Prior Sinusitis Surgery [Number; unit: participants]
  Any Surgery | 32 | 30 | 31 | 93
  Endoscopic sinus surgery | 26 | 28 | 30 | 84
  Balloon sinuplasty | 0 | 0 | 1 | 1
  Polypectomy alone | 5 | 2 | 7 | 14
  Other surgery | 7 | 3 | 7 | 17
Other Chronic Sinusitis Treatment History [Number; unit: participants]
  Systemic antibiotic in last 5 years | 19 | 10 | 19 | 48
  Plan to continue on saline lavage during study (decided at baseline visit) | 20 | 15 | 13 | 48
Smoking History [Number; unit: participants]
  Current Cigarette Smoker | 6 | 12 | 4 | 22
  Current Smoker (other forms of tobacco) | 0 | 0 | 0 | 0
Sinus Imaging in last year [Count of Participants; unit: Participants]
  CT Scans: 0 | 31 | 25 | 32 | 88
  CT Scans: 1 | 41 | 46 | 41 | 128
  CT Scans: 2 | 2 | 2 | 1 | 5
  CT Scans: 3 | 1 | 0 | 0 | 1
  MRI Scans: 0 | 71 | 73 | 71 | 215
  MRI Scans: 1 | 4 | 0 | 3 | 7
  MRI Scans: 2 | 0 | 0 | 0 | 0
  MRI Scans: 3 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Symptoms as Measured by a Composite Score for Each Symptom of Nasal Congestion, Facial Pain or Pressure Sensation, and Nasal Discharge (Anterior and/or Posterior) at the End of Week 4
Description: Change from baseline to the end of Week 4 in average total instantaneous AM scores (evaluation of symptom severity immediately preceding the time of scoring) for each symptom: nasal congestion, nasal discharge (anterior and/or posterior), facial pain/pressure sensation. Baseline scores are the averaged total instantaneous AM scores over the last 7 days of the single blind run in period, and the end of Week 4, scores are averaged over the 7 days from the subject diary. Range of scores for each nasal symptom is 0= none, 1 = mild, 2 = moderate, 3 = severe. Composite score is a sum of the 3 symptom scores and will range from 0 to 9.
Time Frame: 4 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale | -0.81 (0.202) | -1.54 (0.204) | -1.74 (0.204)

2. Primary Outcome: Change From Baseline to Week 24/Early Termination (ET) in the Average Percent of the Volume Opacified (APOV) in the Ethmoid and Maxillary Sinuses.
Description: Change from baseline to Week 24/ET in the average percent of ethmoid and maxillary sinus volume opacified as measured by CT. Percent volume opacified can range from 0% to 100%. Outcome measure is the percentage change from percent opacification at baseline to percent opacification at Week 24; therefore, change in opacification volume can range from -100% to 100%. For example, if Baseline opacification was 68.22% and Week 24 opacification was 66.11%, then the change would be reported as -2.11%.
Time Frame: Baseline, Week 24
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percentage of opacification
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
percentage of opacification | 1.19 (1.740) | -7.00 (1.725) | -5.14 (1.742)

3. Secondary Outcome: Change From Baseline to Week 4 in Each of the 4 Individual Cardinal Chronic Rhinosinusitis (CRS) Symptoms (AM, Instantaneous).
Description: The 4 individual CRS symptoms are: congestion, facial pain or pressure sensation, nasal discharge (anterior and/or posterior), and sense of smell. Range of scores for each nasal symptom is 0= none, 1 = mild, 2 = moderate, 3 = severe. The scores at baseline and week 4 are calculated by averaging the score reported for the individual symptom over 7 days prior to the timepoint. The value provided in the results is calculated by subtracting the score at Week 4 from the score at Baseline; therefore, scores reported here can range from -3 to 3.
Time Frame: Baseline, Week 4
Population: Full analysis set.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale
  Congestion/Obstruction | -0.26 (0.076) | -0.60 (0.077) | -0.70 (0.077)
  Nasal Discharge | -0.27 (0.076) | -0.52 (0.076) | -0.55 (0.077)
  Facial Pain/Pressure | -0.28 (0.080) | -0.44 (0.081) | -0.51 (0.081)
  Sense of Smell | -0.13 (0.066) | -0.24 (0.067) | -0.36 (0.067)

4. Secondary Outcome: Time to First Acute Exacerbation of Chronic Sinusitis
Description: Comparing the distribution of time to first acute exacerbation of chronic sinusitis across treatment groups. An exacerbation of chronic sinusitis is defined as a worsening of symptoms that requires escalation of treatment.
Time Frame: 24 Weeks
Population: Full analysis set.
Measure: Mean (Standard Error); unit: Weeks
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
Weeks | 9.83 (0.215) | 5.00 (0) | 8.04 (0.131)

5. Secondary Outcome: Change From Baseline to Defined Timepoints - Subject Symptoms and Functioning as Measured by the Sinonasal Outcome Test - 22-item (SNOT-22) Total Score and Sub Domains
Description: The SNOT-22 is a subject-completed questionnaire that consists of 22 symptoms and social/emotional consequences of their nasal disorder across several domains including: rhinologic, extra-nasal rhinologic, ear/facial pain, psychological dysfunction, and sleep dysfunction. Total scores range from 0-110. The score range for each domain are as follows: Rhinologic: 0-30; Extra-nasal rhinologic: 0-15; Ear/facial: 0-25; Psychological dysfunction: 0-35; Sleep dysfunction: 0-25. Each item is rated as follows: 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be, and total scores are calculated by adding scores together. The values reported here are calculated by subtracting the score reported at baseline from the score reported at Week 24 and, therefore, can range from the negative maximum score value to the positive maximum score value.
Time Frame: 24 Weeks
Population: Full analysis set.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale
  Total Score | -8.72 (2.186) | -19.45 (2.197) | -15.54 (2.219)
  Rhinologic Symptoms Domain Score | -2.47 (0.649) | -5.25 (0.653) | -4.77 (0.656)
  Extra-Nasal Rhinologic Symptoms Domain Score | -1.61 (0.411) | -2.84 (0.413) | -2.45 (0.415)
  Ear/Facial Symptoms Domain Score | -1.31 (0.613) | -4.45 (0.616) | -3.18 (0.619)
  Psychological Dysfunction Domain Score | -1.80 (0.951) | -5.81 (0.955) | -4.16 (0.965)
  Sleep Dysfunction Domain Score | -1.77 (0.620) | -4.84 (0.622) | -3.61 (0.626)

6. Secondary Outcome: Change From Baseline to Week 8 and 12 in Composite Symptom Score (Congestion, Facial Pain or Pressure Sensation, and Nasal Discharge) for the Total Population and Patients With and Without Previous Sinus Surgery.
Description: Change from baseline in average total instantaneous AM scores (evaluation of symptom severity immediately preceding the time of scoring) for each symptom: nasal congestion, nasal discharge (anterior and/or posterior), facial pain/pressure sensation. Range of scores for each symptom is 0=none, 1=mild, 2=moderate, 3=severe. The composite score is the sum of the 3 symptom scores and will range from 0-9. Scores reported at each timepoint are the averaged total instantaneous AM scores over the last 7 days before the given timepoint. The values presented here are calculated by subtracting the score at Baseline from Week 8 and Week 12, respectively.
Time Frame: 8 weeks, 12 weeks.
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale
  Week 8 Change Total Population | -1.20 (0.210) | -2.02 (0.212) | -2.19 (0.212)
  Week 12 Change Total Population | -1.55 (0.220) | -2.47 (0.223) | -2.60 (0.223)
  Week 8 Change With Prior Surgery Population: number analyzed (Participants) | 27 | 25 | 26
  Week 8 Change With Prior Surgery Population | -1.28 (0.347) | -2.28 (0.355) | -1.95 (0.355)
  Week 12 Change With Prior Surgery Population: number analyzed (Participants) | 27 | 25 | 26
  Week 12 Change With Prior Surgery Population | -1.58 (0.361) | -2.76 (0.379) | -2.36 (0.375)
  Week 8 Change Without Prior Surgery Population: number analyzed (Participants) | 48 | 47 | 47
  Week 8 Change Without Prior Surgery Population | -1.13 (0.263) | -1.86 (0.260) | -2.28 (0.260)
  Week 12 Change Without Prior Surgery Population: number analyzed (Participants) | 48 | 47 | 47
  Week 12 Change Without Prior Surgery Population | -1.51 (0.276) | -2.30 (0.273) | -2.70 (0.274)

7. Secondary Outcome: Change From Baseline to Weeks 8 and 12 in Nasal Congestion Measured by Instantaneous Morning (AM) and Evening (PM) Diary Symptom Scores
Description: Subjects will report instantaneous (evaluation of symptom severity immediately preceding the time of scoring) symptoms. The Nasal Symptom Scale scores as 0=none, 1=mild-symptoms clearly present but minimal awareness, and easily tolerated, 2= moderate - definite awareness of symptoms that is bothersome but tolerable, 3 = severe - symptoms that are hard to tolerate, cause interference with activities or daily living.
Time Frame: 8 Weeks; 12 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale
  Change in AM Score - Week 8 | -0.40 (0.078) | -0.76 (0.079) | -0.84 (0.079)
  Change in PM Score - Week 8 | -0.35 (0.081) | -0.69 (0.082) | -0.75 (0.082)
  Change in AM Score - Week 12 | -0.52 (0.081) | -0.88 (0.082) | -0.97 (0.082)
  Change in PM Score - Week 12 | -0.50 (0.080) | -0.85 (0.081) | -0.91 (0.082)

8. Secondary Outcome: Change From Baseline to Weeks 8 and 12 in Nasal Discharge (Anterior and/or Posterior) Measured by Instantaneous AM and PM Diary Symptom Scores
Description: Subjects will report instantaneous (evaluation of symptom severity immediately preceding the time of scoring) scores. The Nasal Symptom Scale scores as 0=none, 1=mild-symptoms clearly present but minimal awareness, and easily tolerated, 2= moderate - definite awareness of symptoms that is bothersome but tolerable, 3 = severe - symptoms that are hard to tolerate, cause interference with activities or daily living
Time Frame: Baseline, Week 8, Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale
  Change in AM Score - Week 8 | -0.39 (0.080) | -0.63 (0.080) | -0.68 (0.080)
  Change in PM Score - Week 8 | -0.35 (0.081) | -0.66 (0.082) | -0.68 (0.082)
  Change in AM Score - Week 12 | -0.49 (0.085) | -0.83 (0.086) | -0.85 (0.086)
  Change in PM Score - Week 12 | -0.51 (0.085) | -0.83 (0.086) | -0.86 (0.087)

9. Secondary Outcome: Change From Baseline to Weeks 8 and 12 in Facial Pain or Pressure Sensation Measured by Instantaneous AM and PM Diary Symptom Scores
Description: as for outcome 7
Time Frame: Baseline, Week 8, Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale
  Change in AM Score - Week 8 | -0.41 (0.084) | -0.63 (0.085) | -0.67 (0.085)
  Change in PM Score - Week 8 | -0.41 (0.085) | -0.66 (0.086) | -0.70 (0.086)
  Change in AM Score - Week 12 | -0.55 (0.089) | -0.77 (0.090) | -0.78 (0.091)
  Change in PM Score - Week 12 | -0.53 (0.089) | -0.77 (0.091) | -0.78 (0.091)

10. Secondary Outcome: Change From Baseline to Weeks 8 and 12 in Sense of Smell Scores Measured by Instantaneous AM and PM Diary Symptom Scores
Description: Subjects will report instantaneous (evaluation of symptom severity immediately preceding the time of scoring) symptoms. The sense of smell scored as 0= normal, 1=slightly impaired, 2=moderately impaired, 3=absent.
Time Frame: Baseline, Week 8, Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale
  Change in AM Score - Week 8 | -0.18 (0.082) | -0.39 (0.083) | -0.55 (0.083)
  Change in PM Score - Week 8 | -0.13 (0.081) | -0.35 (0.082) | -0.51 (0.082)
  Change in AM Score - Week 12 | -0.32 (0.086) | -0.49 (0.087) | -0.63 (0.087)
  Change in PM Score - Week 12 | -0.29 (0.085) | -0.46 (0.086) | -0.55 (0.086)

11. Secondary Outcome: Change From Baseline to Week 24/ET in the Average Percent of the Volume Opacified in the Ethmoid and Maxillary Sinuses for Patients With and Without Previous Sinus Surgery
Description: Change from Baseline to Week 24/ET in the average percent of ethmoid and maxillary sinus volume opacified as measured by CT for subgroups in patients without and without previous sinus surgery. Percent volume opacified of the combined ethmoid and maxillary sinuses can range from 0% to 100%. Outcome measure is percentage change from percent opacification at baseline to percent opacification at Week 24; therefore, change in opacification volume can range from -100% to 100%. For example, if Baseline opacification was 68.22% and Week 24 opacification was 66.11%, then the change would be reported as -2.11%.
Time Frame: Baseline, Week 24
Population: Full Analysis Set population sizes provided as overall number of participants analyzed. Subgroup population sizes provided with each set of results below.
Measure: Least Squares Mean (Standard Error); unit: percentage of opacification
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
percentage of opacification
  Patients with prior sinus surgery: number analyzed (Participants) | 27 | 25 | 26
  Patients with prior sinus surgery | 3.89 (2.882) | -5.86 (2.862) | -6.73 (2.873)
  Patients without prior sinus surgery: number analyzed (Participants) | 48 | 47 | 47
  Patients without prior sinus surgery | -0.53 (2.118) | -7.83 (2.129) | -4.50 (2.166)

12. Secondary Outcome: Change From Baseline to Week 24/ET in the Lund-Mackay Staging System Total Score
Description: Lund-Mackay Staging System: Lund-Mackay (LM) system (Lund and Mackay, 1993) assigns to each of 10 sinus cavities (left and right maxillary, anterior ethmoid, posterior ethmoid, sphenoid, and frontal) a score of 0 (no opacification), 1 (partial opacification), or 2 (total opacification), plus a 0-2 score for each of the left and right ostiomeatal complex (OMC). The total LM score for a CT scan ranges from 0-24.
Time Frame: Baseline, Week 24
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale | 0.77 (0.332) | -0.54 (0.327) | -0.33 (0.329)

13. Secondary Outcome: Change From Baseline to Week24/ET in the Lund-Mackay Staging System Scores for Each Sinus Pair
Description: Lund-Mackay Staging System: Lund-Mackay (LM) system (Lund and Mackay, 1993) assigns to each of 10 sinus cavities (left and right maxillary, anterior ethmoid, posterior ethmoid, sphenoid, and frontal) a score of 0 (no opacification), 1 (partial opacification), or 2 (total opacification).
  Each sinus pair (left and right side) listed below can achieve a total score of 0-4 (sum of 0-2 for each side). The values reported below are calculated by subtracting the total score at baseline from the total score at Visit 6 (week 24).
Time Frame: Baseline, Week 24
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale
  Anterior Ethmoid Pair | 0.17 (0.071) | 0.03 (0.071) | 0.02 (0.071)
  Posterior Ethmoid Pair | 0.11 (0.071) | 0.04 (0.071) | -0.04 (0.071)
  Maxillary Sinus Pair | 0.04 (0.052) | 0.01 (0.049) | 0.09 (0.049)
  Frontal Sinus Pair | 0.11 (0.093) | -0.12 (0.091) | -0.03 (0.092)
  Sphenoid Sinus Pair | 0.19 (0.078) | -0.04 (0.077) | 0.03 (0.078)

14. Secondary Outcome: Change From Baseline to Week 24/ET in the Average Percent of Sinus Volume Occupied by Disease in the Worst Maxillary Sinus, as Measured by CT Scan Assessment.
Description: Percent volume opacified of the worst maxillary sinus can range from 0% to 100%. The outcome measure is the percentage change from percent opacification of the worst maxillary sinus at baseline to the percent opacification of the same maxillary sinus at Week 24; therefore, change in opacification volume can range from -100% to 100%.
Time Frame: Baseline, Week 24
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percentage of opacification
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
percentage of opacification | -5.83 (2.734) | -14.50 (2.708) | -10.21 (2.724)

15. Secondary Outcome: Change From Baseline to Week 24/ET in the Average Percent of Sinus Volume Occupied by Disease in the Worst Ethmoid Sinus, as Measured by CT Scan Assessment.
Description: Percent volume opacified of the worst ethmoid sinus can range from 0% to 100%. The outcome measure is the percentage change from percent opacification of the worst ethmoid sinus at baseline to the percent opacification of the same ethmoid sinus at Week 24; therefore, change in opacification volume can range from -100% to 100%.
Time Frame: 24 weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percentage of opacification
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
percentage of opacification | -2.79 (1.928) | -9.65 (1.920) | -6.82 (1.928)

16. Secondary Outcome: Change From Baseline to Week 24/ET in the Average Percent of Sinus Volume Occupied by Disease in the Worst Sinus Between Maxillary and Ethmoid Sinuses, as Measured by CT Scan Assessment.
Description: Percent volume opacified of the worst sinus can range from 0% to 100%. The outcome measure is the percentage change from percent opacification of the worst sinus at baseline to the percent opacification of the same sinus at Week 24; therefore, change in opacification volume can range from -100% to 100%.
Time Frame: 24 weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percentage of opacification
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
percentage of opacification | -6.07 (2.493) | -14.02 (2.439) | -10.75 (2.448)

17. Secondary Outcome: Change From Baseline to Week24/ET in the Lund-Mackay Staging System Scores for the Ethmoids and Maxillary Sinuses Combined
Description: Lund-Mackay Staging System: Lund-Mackay (LM) system (Lund and Mackay, 1993) assigns to each of 10 sinus cavities (left and right maxillary, anterior ethmoid, posterior ethmoid, sphenoid, and frontal) a score of 0 (no opacification), 1 (partial opacification), or 2 (total opacification), plus a 0-2 score for each of the left and right ostiomeatal complex (OMC).
  The values reported for this outcome are the change in total opacification of the left an dright maxillary and ethmoid sinuses (Visit 6 [Wk 24] score minus Baseline score). Each visit score can range from a total of 0-12 (sum of 0-2 score assigned for each of left and right maxillary, left and right anterior ethmoid, and left and right posterior ethmoid).
Time Frame: 24 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale | 0.34 (0.162) | 0.09 (0.160) | 0.04 (0.160)

18. Secondary Outcome: Change From Baseline to Week 24/ET in the Zinreich Modification of Lund-Mackay Staging System Total Score
Description: Zinreich modified the LM system by creating subdivisions within "partial opacification" and increasing the range of scores to 0-5 based on percent opacification: 0 = 0%, 1 = 1%-25%, 2 = 26%-50%, 3 = 51%-75%, 4 = 76%- 99%, and 5 = 100% for each each of 10 sinus cavities (left and right maxillary, anterior ethmoid, posterior ethmoid, sphenoid, and frontal). Total score ranges from 0 to 50.
Time Frame: Baseline, Week 24
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale | 0.73 (0.815) | -2.44 (0.806) | -1.45 (0.816)

19. Secondary Outcome: Change From Baseline to Week 24/ET in the Zinreich Modification of Lund-Mackay Staging System for the Sinus Pairs.
Description: Zinreich Modification of the Lund-Mackay Staging System:
  Zinreich modified the LM system by creating subdivisions within "partial opacification" and increasing the range of scores to 0-5 based on percent opacification: 0 = 0%, 1 = 1%-25%, 2 = 26%-50%, 3 = 51%-75%, 4 = 76%- 99%, and 5 = 100%. Each of the following sinus pairs can achieve a total score of 0-10 (sum of score on each left and right side): anterior ethmoids, posterior ethmoids, maxillary sinuses, frontal sinuses, sphenoid sinuses.
  The values reported for this outcome are calculated by subtracting the score at baseline from the score at Visit 6 (Wk 24).
Time Frame: Baseline, Week 24
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale
  Anterior Ethmoid Sinus Pair | 0.18 (0.218) | -0.73 (0.215) | -0.48 (0.217)
  Posterior Ethmoid Sinus Pair | 0.18 (0.239) | -0.54 (0.234) | -0.41 (0.236)
  Maxillary Sinus Pair | 0.17 (0.200) | -0.54 (0.200) | -0.36 (0.202)
  Frontal Sinus Pair | 0.11 (0.250) | -0.37 (0.245) | 0.00 (0.246)
  Sphenoid Sinus Pair | 0.46 (0.249) | -0.32 (0.239) | 0.02 (0.243)

20. Secondary Outcome: Change From Baseline to Week 24/ET in the Zinreich Modification of Lund-Mackay Staging System for Ethmoids and Maxillary Sinuses Combined
Description: Zinreich Modification of the Lund-Mackay Staging System:
  Zinreich modified the LM system by creating subdivisions with "partial opacification" and increasing the range of scores to 0-5 based on percent opacification: 0=0%, 1=1%-25%, 2=26%-50%, 3=51%-75%, 4=76%-99%, and 5=100%. The total score for the combined ethmoids and maxillary sinuses can range from 0-30 (0-5 for each left and right of the anterior ethmoid, posterior ethmoid, and maxillary sinuses). The outcome values presented in the results were determined by subtracting the total score at Baseline from the total score at Week 24.
Time Frame: 24 weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale | 0.51 (0.568) | -1.78 (0.540) | -1.25 (0.546)

21. Secondary Outcome: Change From Baseline to Week 24/ET in the Zinreich Modification of Lund-Mackay Staging System for the Worst Sinus Between Maxillary and Ethmoid Sinuses Among Patient Populations
Description: Zinreich Modification of the Lund-Mackay Staging System:
  Zinreich modified the LM system by creating subdivisions with "partial opacification" and increasing the range of scores to 0-5 based on percent opacification: 0=0%, 1=1%-25%, 2=26%-50%, 3=51%-75%, 4=76%-99%, and 5=100%.
  Data provided for full population and with and without prior sinus surgery subgroups. Number of participants analyzed in the subgroups will be less than the total overall, as these are only portions of the total population.
Time Frame: 24 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale
  Total population | -0.36 (0.137) | -0.93 (0.135) | -0.55 (0.135)
  Prior sinus surgery subgroup: number analyzed (Participants) | 27 | 25 | 26
  Prior sinus surgery subgroup | -0.37 (0.228) | -0.70 (0.223) | -0.64 (0.225)
  Without prior sinus surgery subgroup: number analyzed (Participants) | 48 | 47 | 47
  Without prior sinus surgery subgroup | -0.37 (0.165) | -1.06 (0.167) | -0.52 (0.168)

22. Secondary Outcome: Change in Sleep Quality as Measured by the Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI is a validated, self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate 7 "component" scores (each ranging between 0 and 3): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these 7 components yields 1 global score ranging between 0 and 21. Higher values represent a worse outcome.
Time Frame: 12 Weeks, 24 Weeks
Population: Full analysis set.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale
  Week 12 | -0.27 (0.306) | -1.18 (0.310) | -1.12 (0.307)
  Week 24 | -0.33 (0.293) | -2.01 (0.298) | -1.08 (0.295)

23. Secondary Outcome: Change in Overall Health From Baseline to Week 4 and Week 24/ET as Measured by the Percent of Subjects Improved as Indicated by the Patient Global Impression of Change (PGIC)
Description: Global impression of change will be assessed using a subject-completed PGIC scale range: 1 - Very much improved, 2 - Much improved, 3 - Minimally improved, 4 - No change, 5 - Minimally worse, 6 - Much worse, 7 - Very much worse. Values provided for this outcome measure are the percentage of subjects reporting a score of 1 - Very much improved, 2 - Much improved, or 3 - Minimally improved at each timepoint.
Time Frame: Week 4, Week 24
Population: Full analysis set provided as overall number of participants. Number analyzed at each timepoint is the total number of responders at that timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
Participants
  Week 4: number analyzed (Participants) | 72 | 71 | 71
  Week 4 | 37 | 47 | 56
  Week 24: number analyzed (Participants) | 69 | 70 | 69
  Week 24 | 42 | 59 | 63

24. Secondary Outcome: Change in Baseline to Week 24/ET as Measured by the Short-Form 36 Health Survey, Version 2 (SF-36v2)
Description: The SF-36v2 is a multipurpose, 36-item subject-completed validated questionnaire that measures 8 domains of health: physical functioning, role limitations due to physical health (RP), bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. The SF-36v2 survey with a 4-week recall will be used. It yields scale scores for each of these 8 health domains , each of which is scored from 0 to 100. Higher scores indicate a better health status, with 100 representing the highest level of functioning possible.
Time Frame: 24 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale
  Physical Functioning Score | 0.54 (1.012) | 3.46 (1.023) | 2.24 (1.043)
  Role Physical Score | 0.18 (1.018) | 5.02 (1.029) | 3.73 (1.049)
  Bodily Pain Score | 2.46 (1.193) | 5.74 (1.205) | 3.54 (1.223)
  General Health Score | -0.20 (1.010) | 4.71 (1.025) | 2.78 (1.037)
  Vitality Score | 0.35 (1.120) | 4.59 (1.129) | 3.98 (1.157)
  Social Functioning Score | -0.11 (1.173) | 4.70 (1.186) | 1.58 (1.204)
  Role Emotional Score | -0.77 (1.133) | 2.23 (1.147) | 0.42 (1.167)
  Mental Health score | -1.70 (1.100) | 2.26 (1.112) | 1.23 (1.138)

25. Secondary Outcome: Change in the 36-Item Short Form Health Survey Version 2 (SF-36v2) Mental Component Score (MCS).
Description: Change from baseline to Week 24/ET on the MCS of the 36-Item Short Form Health Survey version 2 (SF-36v2). The SF-36v2 is a multipurpose, scaled, 36-item, subject-completed validated questionnaire. The scale range is from 0-100. A lower score means more disability and a higher score means less disability. Result values are calculated by subtracting the score reported at Week 24 from the score reported at Baseline.
Time Frame: 24 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale | -0.82 (0.888) | 2.25 (0.895) | 1.17 (0.913)

26. Secondary Outcome: Change in the SF-36v2 Physical Component Score (PCS)
Description: Change from baseline to Week 24/ET on the PCS of the 36-Item Short Form Health Survey version 2 (SF-36v2). The SF-36v2 is a multipurpose, scaled, 36-item, subject-completed validated questionnaire. The scale range is from 0-100. A lower score means more disability and a higher score means less disability. Result values are calculated by subtracting the score reported at Week 24 from the score reported at Baseline.
Time Frame: 24 Weeks
Population: full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale | 2.12 (0.712) | 5.35 (0.723) | 4.34 (0.738)

27. Secondary Outcome: Change in Depressive Symptoms From Baseline to Week 24/ET as Measured by Change in the Severity of Depression as Measured by the Quick Inventory of Depression Symptomatology (QIDS)
Description: The 16-item QIDS (Rush et al. 2003) is designed to assess the severity of depressive symptoms. The QIDS is available in a self-rated version and assesses all the criterion symptom domains designated by the American Psychiatry Association Diagnostic and Statistical Manual of Mental Disorders - 5th edition to diagnose a major depressive episode. The 7-day period prior to assessment is the usual time frame for assessing symptom severity. Scores range from 0 to 27, where higher scores indicate a worse outcome.
Time Frame: 24 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale | -0.23 (0.306) | -0.74 (0.308) | -0.20 (0.312)

28. Secondary Outcome: Severity of Depression at Week 24 as Measured by the Quick Inventory of Depression Symptomatology (QIDS)
Description: The 16-item QIDS (Rush et al. 2003) is designed to assess the severity of depressive symptoms. The QIDS is available in a self-rated version and assesses all the criterion symptom domains designated by the American Psychiatry Association Diagnostic and Statistical Manual of Mental Disorders - 5th edition to diagnose a major depressive episode. The 7-day period prior to assessment is the usual time frame for assessing symptom severity. Scores range from 0 to 27, where higher scores indicate a worse outcome. Results reported for this outcome measure are the
Time Frame: 24 Weeks
Population: Overall number of participants analyzed is the total number of responders at Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 69 | 71 | 69
Participants
  No depression | 52 | 55 | 51
  Mild depression | 15 | 12 | 15
  Moderate depression | 0 | 4 | 2
  Severe depression | 0 | 0 | 1
  Very severe depression | 2 | 0 | 0

29. Secondary Outcome: Change in Olfactory Impairment From Baseline to Week 24/ET as Measured by the Smell Identification Test (SIT)™
Description: The SIT is a test comprised of 4 booklets each containing 10 microencapsulated (scratch and sniff) odors. Forced choice response alternatives accompany each test item. Each correct response is assigned a score of 1 and incorrect responses are assigned a score of 0. The total score is calculated by summing the scores of each individual odor for a total possible score ranging from 0-40. The higher the score, the better the individual's sense of smell. The test provides an absolute indication of smell loss (anosmia; mild, moderate or sever hyposmia) as well as an index to detect malingering.
Time Frame: 24 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale | 0.23 (0.954) | 2.63 (0.959) | 0.70 (0.972)

30. Secondary Outcome: Change in Baseline to Week 24/ET as Measured by the Euroqol 5-dimension (EQ-5D) Instrument
Description: The EQ-5D consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The outcome measured for this study was the EQ VAS, which records the subject's self-rated health on a vertical visual analogue scale, where the endpoints are labelled "The best health you can imagine" and "The worst health you can imagine". The VAS can be used as a quantitative measure of health outcome that reflects the subject's own judgement. VAS scores range from 0 (worst health you can imagine) to 100 (best health you can imagine).
Time Frame: 24 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale | 2.10 (1.889) | 9.67 (1.880) | 7.30 (1.891)

31. Secondary Outcome: Change in Baseline to Week 24/ET as Measured by the Short-Form 6-Dimension (SF-6D) Instrument
Description: The SF-6D is a single health state index derived from the 11 items from the SF-36v2. SF-6D scores range from 0 (worst health state) to 1 (best health state). The values provided in the outcome data are calculated by subtracting the score reported at baseline from the score reported at Visit 6 (Week 24).
Time Frame: 24 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 72 | 73
score on a scale | 0.00 (0.016) | 0.06 (0.016) | 0.05 (0.016)

32. Secondary Outcome: Percentage of Subjects Indicating That They Are Willing to Consider Sinus Surgery at Baseline and Week 24
Description: Percentage of subjects indicating that they are willing to consider Sinus Surgery. This is a comparison of health economic measures and data was obtained by direct questioning of the subjects during study visits.
Time Frame: Baseline, Week 24
Population: Overall number of participants analyzed is total number of responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 70 | 69 | 69
Participants
  Baseline | 38 | 40 | 38
  Week 24 | 35 | 36 | 33

33. Secondary Outcome: Percentage of Subjects Who Meet the Minimal Objective Criteria for Surgical Intervention at Baseline and Week 24.
Description: Percentage of subjects who meet the minimal objective criteria for surgical intervention based on completion of a surgical intervention assessment questionnaire for the investigator.
Time Frame: Baseline, Week 24
Population: Overall number of participants analyzed is total number of responders in each treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 66 | 70 | 69
Participants
  Baseline | 15 | 6 | 15
  Week 24 | 14 | 3 | 10

34. Secondary Outcome: Percentage of Subjects Approved for Surgery Who no Longer Elect to Undergo a Surgery
Description: Outcome value presented here is the percent of subjects who are approved for surgery but no longer elect to undergo a surgery. Number of participants analyzed indicates the total number of participants for whom this analysis was completed.
Time Frame: Week 24
Population: Total number of responders in each treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 70 | 69 | 69
Participants | 35 | 33 | 36

35. Other Pre Specified Outcome: Evaluation of Safety by Recording the Severity of Adverse Events (AEs)
Description: Assessment of safety by measuring severity of AEs using scale with 1=mild, 2=moderate, 3=severe
Time Frame: 24 Weeks
Population: Safety analysis set. Values provided for this outcome are the count of subjects with at least 1 AE in each category.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 73 | 74
Participants
  Mild | 13 | 15 | 22
  Moderate | 17 | 8 | 19
  Severe | 1 | 1 | 2

36. Other Pre Specified Outcome: Evaluation of Safety-Nasal Examination
Description: Assessed in nasal examination worksheet which includes recording the presence of any epistaxis, septal erosion/perforation, ulceration/erosion of area other than septum.
Time Frame: 24 Weeks
Population: Safety analysis set. Overall number analyzed is the total number of responders in each treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 71 | 71 | 72
Participants
  Epistaxis: None | 71 | 70 | 68
  Epistaxis: Present | 0 | 1 | 4
  Septal erosion/perforation: None | 70 | 71 | 70
  Septal erosion/perforation: Present | 1 | 0 | 2
  Ulceration/Erosion: None | 71 | 71 | 72
  Ulceration/Erosion: Present | 0 | 0 | 0
  Mucosal candidiasis: None | 71 | 71 | 72
  Mucosal candidiasis: Present | 0 | 0 | 0

37. Other Pre Specified Outcome: Evaluation of Safety Measuring Vital Signs- Blood Pressure
Description: Includes systolic and diastolic blood pressure measurements in millimeter of mercury (mmHg)
Time Frame: 24 Weeks
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 73 | 74
mmHg
  Systolic Blood Pressure | 126.2 (11.30) | 124.0 (13.26) | 126.9 (11.94)
  Diastolic Blood Pressure | 78.1 (8.29) | 76.5 (7.88) | 78.5 (7.69)

38. Other Pre Specified Outcome: Evaluation of Safety Measuring Vital Signs- Pulse
Description: Measure pulse in beats per minute (bpm)
Time Frame: 24 Weeks
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 73 | 74
beats per minute | 73.7 (7.37) | 74.1 (6.76) | 72.1 (8.18)

39. Other Pre Specified Outcome: Evaluation of Safety Measuring Vital Signs- Weight
Description: Assessment of safety from physical examination-weight measured in kg or lb
Time Frame: 24 Weeks
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 73 | 74
kg | 77.86 (16.527) | 76.30 (15.250) | 81.14 (20.091)

40. Other Pre Specified Outcome: Evaluation of Safety - Monitoring Concomitant Medication Usage
Description: Assessment for safety from the collection of information for concomitant medications usage. Top 5 reported con-meds by therapeutic class are listed for this outcome.
Time Frame: 24 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
Number analyzed (Participants) | 75 | 73 | 74
Participants
  Other Nasal Preparations (includes sodium chloride and sea water) | 22 | 15 | 15
  Adrenergics in combination with corticosteroids or other drugs | 15 | 9 | 19
  Glucocorticoids | 11 | 9 | 7
  Selective Beta-2-adrenoreceptor Agonists | 11 | 4 | 8
  HMG-CoA Reductase Inhibitors | 8 | 7 | 9

ADVERSE EVENTS:
Time Frame: Pretreatment (Screening/Run-in) period to end of treatment (Week 24)
Description: Total number of participants at risk is defined by the Safety Analysis Set, which is all enrolled/randomized subjects who received at least 1 dose of randomized study treatment. The number of participants in the Safety Analysis Set differs from the Full Analysis Set (total population analyzed for the outcome measures) due to two participants who discontinued the study, meeting the criteria for inclusion in the Safety Analysis Set but not the Full Analysis Set.
Arm/Group | Placebo | OPN-375 186 μg BID | OPN-375 372 μg BID
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/73 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/75 | 1/73 | 4/74
Other Adverse Events (participants affected / at risk) | 31/75 | 17/73 | 43/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=75) | OPN-375 186 μg BID (N=73) | OPN-375 372 μg BID (N=74)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | OPN-375 186 μg BID (N=73) | OPN-375 372 μg BID (N=74)
Cataract nuclear (Eye disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 2
COVID-19 (Infections and infestations) | 2 | 3 | 7
Nasopharyngitis (Infections and infestations) | 5 | 3 | 4
Chronic Sinusitis (Infections and infestations) | 5 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1
Influenza (Infections and infestations) | 0 | 2 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Vaccination complication (Injury, poisoning and procedural complications) | 2 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Headache (Nervous system disorders) | 6 | 2 | 7
Sinus headache (Nervous system disorders) | 0 | 0 | 2
Depression (Psychiatric disorders) | 1 | 0 | 3
Persistent depressive disorder (Psychiatric disorders) | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 7
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT03960580/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT03960580/SAP_001.pdf